CLINICAL TRIAL: NCT01122485
Title: For an 8-week, Single Center, Randomized, Double Blind, Placebo Controlled Exploratory Clinical Study to Assess the Efficacy, Dose Response and Safety of PG201 Tablet in Patients With Osteoarthritis
Brief Title: Efficacy and Safety Study of PG201 Tablet in Patients With Osteoarthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This product was licensed to another Korean company, no study data is available.
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG201-PT-001
Record Dates: First submitted 2010-05-06; First posted 2010-05-13 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — herbal extract PG201

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose group (Experimental): two tablets per dose (one tablet of investigational drug and one tablet of placebo)
  Interventions: Other: PG201
- High dose group (Experimental): two tablets per dose (two tablets of investigational drug)
  Interventions: Other: PG201
- Control group (Placebo Comparator): two tablets per dose (two tablets of placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: PG201 — two tablets
  Other Names: Botanical drug
  Arms: High dose group; Low dose group
Other: Placebo — two tablets
  Other Names: control drug(placebo)
  Arms: Control group

SUMMARY:
The objective of this study was to explore the efficacy, dose-response and safety of PG201 tablet in Korean patients with osteoarthritis.

DETAILED DESCRIPTION:
In this study, the PG201 extract, the study drug, was administered twice daily after a meal to two investigational groups, the lower-dose group and the higher-dose group. The efficacy of each of dose group was compared to that of the control group to determine if there was a statistically significant difference between the investigational groups and the placebo group. In addition, the efficacy between the lower dose group and the high dose group was also compared to determine if there was a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥40 and ≤ 75 years of age
* For a woman, she should meet one of the following criteria to be eligible for the study: i) A woman of no childbearing potential ii) As for a woman of childbearing potential, she should have a negative pregnancy test result at screening and baseline/randomization
* Patients should be able and willing to provide the written informed consent.
* Patients should be able to read and understand the information provided for the study and be able to record the information requested by the study.
* Patients who meet the American College of Rheumatology clinical plus radiographic classification criteria for idiopathic osteoarthritis of the knee, which are defined as follow: a patient who had knee pain and radiographically diagnosed osteophytes and met at least one of the followings. i) Age> 50 years ii) Morning stiffness for less than 30 minutes iii) Crepitus during movement of the weight-bearing knee
* Patients with symptomatic primary osteoarthritis of the knee at least in the last 3 months prior to screening.
* Patients with severity of grade 2 or 3 according to Kellgren & Lawrence scale based on anteroposterior radiographic evidence of the tibiofemoral joints with osteoarthritis, and who are classified in functional class of I, II or III according to the American Rheumatism Association functional classification.
* Patients who had a score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale question 1 ≤80 mm at screening, a score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale question 1 ≥50 mm at baseline. a decrease in the score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale question 1 at least by 15mm from screening to baseline and a decrease in the patient self-assessed arthritis symptoms scores at least by one point from screening to baseline.
* Patients who received Nonsteroidal antiinflammatory drugs (NSAIDs)/Cyclooxygenase-2 inhibitor for the treatment of arthritis of the knee for at least 5 days a week during 4 weeks prior to screening

Exclusion Criteria:

* Patients with a known hypersensitivity or intolerance to Nonsteroidal antiinflammatory drugs (NSAIDs), aspirin or Cyclooxygenase-2 inhibitor.
* Patients with a clinical or biochemical abnormal finding (excluding any finding related to the investigating disease) at the screening visit, which in the investigator's opinion was considered to be clinically significant or might make safe participation in the study more difficult
* Patients with a history of gastroduodenal perforation and/or occlusion, gastric or duodenal surgery, progressive upper gastrointestinal ulcer within the last 6 months or a history of upper gastrointestinal bleeding (including hematemesis) within the last one year, lower gastrointestinal bleeding within the last one year (excluding hemorrhoid), inflammatory intestinal disease within the last 6 months, coronary artery disease, congestive heart failure or renal artery stenosis, stroke or transient ischemic attack.
* Patients with uncontrollable hypertension
* Patients receiving aspirin therapy (low-dose aspirin in a daily dose of 325mg or less is permitted for prevention of cardiovascular disease).
* Patients receiving anticoagulant drug or antiplatelet drug (excluding low-dose aspirin) or who have a disease associated with hemostatic disorder.
* Patients with any of creatinine, bilirubin, Alanine aminotransferase or Aspartate aminotransferase > 1.5 times the Upper Lange of normal at screening. Patients who have any two or more of bilirubin, Alanine aminotransferase or Aspartate aminotransferase level greater than the Upper Lange of normal will also be excluded.
* Patients with a history of drug or alcohol abuse.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Estimated); Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Pain score on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Day 56

SECONDARY OUTCOMES:
Sub-scale score and total score on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Day 28
The responder index (RI) | Screening, Day 1, Day 28
The change in the quality of life score | Day 1, Day 28
The change in the patient self-assessed overall symptom scores | Screening, Day 1, Day 28
The change in the investigator-assessed overall symptom scores | Screening, Day 1, Day 28
Adverse event, and the presence and incidence of abnormal laboratory | Screening, Day 1, Day 28, Day 56

CONTACTS AND LOCATIONS:
Overall Officials: S.H. Park, M.D., Principal Investigator — Dept. of Rheumatology, Seoul St. Mary's Hospital, The Catholic University of Korea